CLINICAL TRIAL: NCT06959030
Title: An Observational Study on the Safety and Efficacy of Henagliflozin in Chinese Patients With Type 2 Diabetes
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Liang Yuzhen, Director of Endocrinology Department, chief physician, MD, doctoral supervisor, Second Affiliated Hospital of Guangxi Medical University
Other Study IDs: MA-DM-Ⅳ-012
Record Dates: First submitted 2025-04-16; First posted 2025-05-06 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention: Observational Cohort — Observation study

SUMMARY:
An Observational Study on the Safety and Efficacy of Henagliflozin in Chinese Patients with Type 2 Diabetes Primary Research Objective

• To evaluate the safety of Henagliflozin in Chinese patients with type 2 diabetes mellitus (T2DM) in real world.

Exploratory Research Objectives

* 1. Improvement in metabolic parameters: To assess changes in metabolic indicators, including glycated hemoglobin (HbA1c), fasting plasma glucose (FPG), 2-hour postprandial plasma glucose (PPG), blood pressure, and body weight, in T2DM patients treated with Henagliflozin.
* 2. Incidence of specific adverse events: To investigate the occurrence of key adverse events, with a focus on hypovolemia, amputation or amputation risk, fractures, urinary tract infections, genital infections, renal impairment, diabetic ketoacidosis, hepatic dysfunction, and severe hypoglycemia.
* 3. Impact on muscle health: To evaluate changes in muscle health indicators, such as skeletal muscle mass index, lean body mass, and grip strength, in T2DM patients receiving Henagliflozin therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old≤ age ≤ 80 years old;
2. Diagnosed with type 2 diabetes mellitus according to WHO diagnostic criteria, currently receiving or eligible for add-on therapy with Henagliflozin;
3. Voluntarily participate in this study and sign the informed consent form. If the subject does not have the ability to read the informed consent form (e.g., illiterate subjects), a witness is required to witness the informed process and sign the informed consent form.

Exclusion Criteria:

1. Participation in or current enrollment in clinical trials investigating other glucose-lowering medications within 1 month prior to the initiation of this study.
2. Current or history of recurrent urinary tract infections (UTIs) and/or genital infections.
3. Patients judged by the investigator to be unsuitable to participate in this clinical trial, with considerations such as current blood volume status, estimated glomerular filtration rate (eGFR), and other clinical parameters.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chinese Patients with Type 2 Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
incidence of adverse events and serious adverse events during 24 weeks of treatment | 24 weeks

SECONDARY OUTCOMES:
changes of HbA1c (mmol/L) in T2DM patients during treatment with Henagliflozin | 24 weeks
  Exploratory Research Objectives
changes of fasting plasma glucose (FPG) in T2DM patients during treatment with Henagliflozin | 24 weeks
changes of 2-hour postprandial plasma glucose (PPG) in T2DM patients during treatment with Henagliflozin | 24 weeks
changes of blood pressure in T2DM patients during treatment with Henagliflozin | 24 weeks
changes of weight in T2DM patients during treatment with Henagliflozin | 24 weeks
incidence of specific adverse events during 24 weeks of treatment | 24 weeks
  specific adverse events (including abnormal liver function test, urinary tract infection, genital infection, hypovolemia, renal events, serious hypoglycemia events, fractures, diabetic ketoacidosis, amputation caused by adverse events or with amputation risk)
changes of limb skeletal muscle mass index in T2DM patients during treatment with Henagliflozin | 24 weeks
changes of lean body mass in T2DM patients during treatment with Henagliflozin lean body mass | 24 weeks
changes of grip strength in T2DM patients during treatment with Henagliflozin | 24 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The People's Hospital of Beihai, Beihai, Guangxi
  - Guilin Municipal Hospital of Traditional Chinese Medicine, Guilin, Guangxi
  - Nanxishan Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - the Second Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Qingdao Aikangyi Internet Hospital, Qingdao, Shandong

IPD SHARING:
Plan to Share IPD: No